CLINICAL TRIAL: NCT06438120
Title: Chatbot-based Positive Psychology Intervention to Promote Well-being in Caregivers of Children With Autism Spectrum Disorder: A Pilot Feasibility Study
Brief Title: Chatbot-based Positive Psychology Intervention in Caregivers of Children With Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Wendy Zhang Wen, Assistant Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RD/2023/1.20
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Participants will receive chatbot-based positive psychology exercises including positive introduction, personal strengths, using strengths, three good things, gratitude letter/visit, hope and optimism, active/constructive responding, and savoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chatbot group (Experimental): In this group, participants will receive chatbot-based positive psychology intervention.
  Interventions: Behavioral: Chatbot-based positive psychology intervention

INTERVENTIONS:
Behavioral: Chatbot-based positive psychology intervention — Eight positive psychology exercises will be delivered, including positive introduction, personal strengths, using strengths, three good things, gratitude, hope and optimism, active/constructive responding, and savoring.

SUMMARY:
This project aims to evaluate the feasibility and preliminary effectiveness of chatbot-based positive psychology intervention.

DETAILED DESCRIPTION:
According to a World Health Organization report, one in 100 children is diagnosed with Autism Spectrum Disorder (ASD), which is characterized by varying degrees of disability and deviation in social communication and interaction. Half of the parents of children with ASD have reported showing depression and high levels of anxiety. Lower well-being and poor quality-of-life have also been reported. Thus, there is an urgent need to find applicable interventions to reduce depressive symptoms and promote mental health in caregivers of children with ASD.

Positive psychology intervention uses positive psychological skills, such as savoring, gratitude, forgiveness, optimism, personal strength, and attainable goals, to identify meaning and value in life events and to promote positive emotions, cognitions and behaviors. Considering the convenience, low cost and popularity of chatbot, chatbot-based positive psychology intervention will be applied in this study. A pilot feasibility study will be proposed to evaluate the feasibility of chatbot-based positive psychology intervention.

The primary objective is to evaluate the feasibility and preliminary effectiveness of chatbot-based positive psychology intervention in promoting well-being in caregivers of children with ASD (Primary).

The secondary objectives are:

To test if the intervention reduces perceived stress in caregivers of children with ASD; To test if the intervention reduces depressive symptoms of caregivers of children with ASD; To test if the intervention improves quality of life in caregivers of children with ASD.

ELIGIBILITY:
Inclusion criteria:

Primary caregivers

* (i) providing long-term care for the primary-school-age child (6-11 years old) diagnosed with ASD;
* (ii) who are over 18 years old;
* (iii) who have the ability to communicate and read in Chinese;
* (iv) who have at least one mobile phone with an internet connection.

Exclusion criteria:

Primary caregivers

* (i) who participate in a similar psychological intervention within one year;
* (ii) currently on regular psychotropic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The score of feasibility | After the intervention immediately
  Feasibility will be assessed by 2 items modified from the Feasibility of Intervention Measure, and the semi-structured interview will be conducted immediately after the intervention (9-week follow-up). Barriers and facilitators to participant adherence and retention will be discussed to collect feedback. These 2 items will ask participants to evaluate that the Chatbot is implementable and easy to use via a 5-point Likert scale from completely disagree (1) to completely agree (5). The score range is 2 to 10 and higher scores indicate greater feasibility.
Qualitative results of feasibility | After the intervention immediately
  The focus group will be conducted to learn about the barriers and facilitators to participant adherence, and retention will be discussed to collect feedback. The perspectives on potential feasibility, acceptability, facilitators, barriers, priority domains, and suggestions for the Chatbot will be discussed.
The score of well-being | Baseline and after the intervention immediately
  Well-being will be measured by the World Health Organization-5 Well-being Index to evaluate vitality (being active and waking up fresh and rested), being interested in things, and having a pleasant attitude. Each item is scored using a 6-point Likert scale from at no time (0) to all of the time (5). The total score ranges from 0 to 25, with higher scores suggesting better self-perceived well-being.

SECONDARY OUTCOMES:
Perceived Stress | Baseline and after the intervention immediately
  Perceived Stress will be assessed by a 10-item Perceived Stress Scale (PSS-10) with a 5-point Likert scale from never (0) to very often (4). The total score is from 0 to 40 and a higher score reflects a higher level of perceived stress.
Depressive symptoms | Baseline and after the intervention immediately
  Depressive symptoms will be measured by the Patient Health Questionnaire-9 (PHQ-9), which evaluates the frequency of occurrence of main depressive symptoms over the past 2 weeks via a 4-point Likert scale from not at all (0) to nearly every day (3). The total score is from 0 to 27 and the higher scores indicate more severe depressive symptoms.
The score of Quality of life | Baseline and after the intervention immediately
  Quality of life will be measured by the Chinese version of Short Form-8(SF-8), including 8 sub-scales: general health perception, physical function, bodily pain, role limitations due to physical health problems, vitality, role limitations due to emotional problems, social function, and mental health. A norm-based scoring method will be applied to calculate physical summary scores and mental summary scores. The sub-scale score can be represented as T-scores(mean =50, standard deviation =10) and a higher score indicating better QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong